CLINICAL TRIAL: NCT02645630
Title: Effects of Pain, Disability, Widespread Pressure Pain Sensitivity, and Cervicokinesthesia After Cervical Manipulation in Patients With Mechanical Neck Pain
Brief Title: Effects of Pain, Disability and Cervicokinesthesia After Cervical Manipulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, César Fernández-de-las-Peñas, Head Division, Universidad Rey Juan Carlos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: URJC2015-161120155015
Record Dates: First submitted 2015-12-30; First posted 2016-01-05 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-12

CONDITIONS: Neck Pain
Keywords: Cervical spine; Spinal manipulation
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Right Cervical Manipulation (Experimental): Patients assigned to this group will receive a cervical spine manipulation targeting the C3/C4 segment on the right side.
  Interventions: Other: Right Cervical Manipulation
- Left Cervical Manipulation (Experimental): Patients assigned to this group will receive a cervical spine manipulation targeting the C3/C4 segment on the left side.
  Interventions: Other: Left Cervical Manipulation
- Sham Cervical Manipulation (Active Comparator): Patients assigned to this group will receive a sham cervical spine manipulation targeting the C3/C4 segment on both sides. No therapeuthic thrust will be applied.
  Interventions: Other: Sham Cervical Manipulation

INTERVENTIONS:
Other: Right Cervical Manipulation — We will use a high-velocity, mid-range, left rotational force to the right articular pillar of C3, on the right articular pillar of C4 with the patient in supine, with left rotation and right side-bending.
  Arms: Right Cervical Manipulation
Other: Left Cervical Manipulation — We will use a high-velocity, mid-range, left rotational force to the left articular pillar of C3, on the left articular pillar of C4 with the patient in supine, with right rotation and left side-bending.
  Arms: Left Cervical Manipulation
Other: Sham Cervical Manipulation — The sham procedure will simulate C3/C4 manipulation in both sides without any therapeutic thrust
  Arms: Sham Cervical Manipulation

SUMMARY:
Cervical spine manipulation has been found to be effective in patients with mechanical neck pain. Discrepancies exist on the side of manipulation and the placebo effect of this manual intervention. In addition, some authors have proposed that spinal manipulation can alter proprioception of the cervical spine. The aim of this study will be to investigate the effects of cervical spine manipulation on pain, disability, widespread pressure pain sensitivity, and cervicokinethesia in patients with mechanical neck pain.

DETAILED DESCRIPTION:
Cervical spine manipulation has been found to be effective in patients with mechanical neck pain. Discrepancies exist on the side of manipulation and the placebo effect of this manual intervention. In addition, some authors have proposed that spinal manipulation can alter proprioception of the cervical spine. The aim of this study will be to investigate the effects of cervical spine manipulation on pain, disability and cervicokinethesia in patients with mechanical neck pain. Patients will receive cervical spine manipulation in either right or left side of the neck and will be assessed on pain intensity, neck-related disability, widespread pressure pain sensitivity, and cervicokinethesia by an assessor blinded to the allocation group.

ELIGIBILITY:
Inclusion Criteria:

- Generalized neck-shoulder pain with symptoms provoked by neck postures, neck movement, or palpation of the cervical musculature.

Exclusion Criteria:

* any contraindication to manipulation, e.g., positive extension-rotation test;
* whiplash injury;
* previous cervical surgery;
* cervical radiculopathy or myelopathy;
* diagnosis of fibromyalgia syndrome;
* having undergone spinal manipulative therapy in the previous 6 months;
* less than 18 or greater than 65 years of age.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2015-12; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Changes in cervical kinesthetic sense before and after the intervention | Baseline and 15 minutes after the intervention
  The joint position sense error (JPSE) will be calculated to determine cervicokinethesia

SECONDARY OUTCOMES:
Changes in disability before and after the intervention | Baseline and one week after the intervention
  The Neck Disability Index (NDI) will be used to determine neck-related disability
Changes in neck pain intensity before and after the intervention | Baseline and one week after the intervention
  An 11 points numerical pain rate scale (NPRS, 0-10) will be used to assess the intensity of neck pain
Changes in widespread pressure pain sensitivity before and after the intervention | Baseline and 15 minutes after the intervention
  Pressure pain thresholds will be assessed over C5/C6 zygapophyseal joints and the tibialis anterior muscle

CONTACTS AND LOCATIONS:
Overall Officials: CESAR FERNANDEZ-DE-LAS-PEÑAS, PT, PhD, Principal Investigator — Universidad Rey Juan Carlos
Locations (1):
- Cesar Fernandez-de-Las-Peñas, Alcorcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No